CLINICAL TRIAL: NCT04066387
Title: Characteristics and Prognosis of Patients With Critical Ischemia at High Risk of Amputation Managed by Endovascular Bypass: a Retrospective Study of 15 Patients
Acronym: Pontage
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: Pontage
Record Dates: First submitted 2019-08-22; First posted 2019-08-26 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2019-10

CONDITIONS: Limb Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Obliterative arterial disease of the lower limbs (AOMI) is associated with a high risk of cardiovascular events, with a linear relationship between a fall in the systolic pressure index and a risk of cardiovascular morbidity and mortality. Critical ischemia is the most severe stage of AOMI, associated with decubitus pain and / or foot ulceration. The severity of this arterial involvement involves functional prognosis of the lower limb with a high risk of amputation, as well as the patient's vital prognosis. In these patients, the rate of amputation and mortality at 1 year can reach 20%. Consequently, the goal of management in a multidisciplinary setting is threefold: the treatment of pain, improvement of the functional prognosis and improvement of the patient's vital prognosis. Revascularization should be attempted as often as possible for the purpose of limb salvage and improvement of patient survival.

In the vascular medicine department, the indication and modalities of the revascularization procedure are discussed at a multidisciplinary consultation meeting. The medical-radiological-surgical expertise takes into consideration the patient's terrain and comorbidities and the technical possibilities according to the arterial damage. With the modernization and development of endovascular equipment dedicated to the hamstrings, the interventional radiology techniques in the management of critical ischemia allow the treatment of one or more arterial axes as well as a very distal revascularization in the arteries. foot with a lower morbidity-mortality compared to surgery, especially in the most fragile patients. Since 2013, the endovascular revascularization procedures performed by the interventional radiology team have been an integral part of the management of patients with critical ischemia hospitalized in the vascular medicine department.

In patients with critical ischemia at high risk of major amputation and without the option of traditional endovascular or surgical revascularization, an endovascular revascularization technique for leg rescue is discussed as a last resort in multidisciplinary staff. This technique, performed by the interventional radiology team (MDP and GA), consists of an extra-anatomic endovascular femoro-popliteal bypass. We wish to describe the limb salvage rate and the preservation of autonomy in the 15 patients treated with this revascularization technique since 2013 in the vascular medicine department of the GHPSJ.

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age ≥ 18 years
* Patient with critical ischemia at high risk of amputation without the option of "traditional" surgical or endovascular revascularization after multidisciplinary staff discussion
* Patient treated by the non-surgical technique called "endovascular bypass"
* Patient with preserved autonomy

Exclusion Criteria:

* Patient presenting a loss of autonomy, genu flessum analgesic
* Patient with a contraindication to antithrombotic therapy
* Patient with infectious complications of life-threatening ischemic wounds
* Patient under tutorship or curatorship
* Patient deprived of liberty
* Patient opposing the use of his data for this research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - Patient with critical ischemia at high risk of amputation without the option of "traditional" surgical or endovascular revascularization after multidisciplinary staff discussion, treated by the non-surgical technique called "endovascular bypass"
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Member rescue rate | year 1
  This outcome measure the member rescue rate.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra P YANNOUTSOS, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided